CLINICAL TRIAL: NCT07080541
Title: Natural-Based Multicomponent Intervention to Promote Quality of Life and Healthy Habits on Children and Adolescents: Protocol for a Randomized Controlled Trial
Brief Title: Protocol for a Natural-Based Intervention to Promote Quality of Life and Healthy Habits on Children and Adolescents.
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Extremadura (Other)
Responsible Party: Principal Investigator, Noelia Mayordomo, PhD Student/Substitute professor, Universidad de Extremadura
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Health Services Research
Other Study IDs: 139//2024
Record Dates: First submitted 2025-05-26; First posted 2025-07-23 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: Life Quality; Physical Activities; Life Style, Healthy; Life Style Modification
Keywords: physical activity; physical literacy; quality of life; natural environment; nature
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Physical literacy information (Experimental): Participants in the technology experimental group received physical literacy and life satisfaction information prior to the adventure activities via social media.
  Interventions: Other: Physical literacy and life satisfaction
- Analogic information (Experimental): Participants in the analogic experimental group received physical literacy and life satisfaction information prior to the adventure activities using paper sheets.
  Interventions: Other: Analogic information
- Participants physical activity intervention (no information) (No Intervention): Participants in the analogic experimental group received physical literacy and life satisfaction information prior to the adventure activities using paper sheets.

INTERVENTIONS:
Other: Physical literacy and life satisfaction — Participants in the technology experimental group will engage in physical activity in nature while being exposed to information pills on physical literacy and the importance of physical activity in health to improve quality of life and life satisfaction via social media
  Arms: Physical literacy information
Other: Analogic information — Participants in the analogic experimental group will engage in physical activity in nature while being exposed to information pills on physical literacy and the importance of physical activity in health to improve quality of life and life satisfaction via paper sheets.
  Arms: Analogic information

SUMMARY:
In current society, physical activity practices show a decreasing trend, together with a low perception of life quality. In addition, urban overcrowding has led to disconnection from the natural environment, causing the benefits that this context offers to be lost, especially for children and adolescents. Physical literacy is an approach to physical activity that encompasses more than just individual physical skills. It emphasises the importance of performing physical activity on a regular basis as part of daily life, encompassing bodily expression and understanding, as well as self-confidence and motivation, making it a factor that contributes to quality of life. Although research shows a correlation between physical literacy and life satisfaction, there is no research on other variables, such as the impact of green spaces in this correlation. This study aimed to present the rationale and methods of a randomized controlled trial in green spaces for children and adolescents aged 8 to 18 to evaluate the efficacy of a nature-based intervention designed to promote healthy habits through physical literacy and quality of life through life satisfaction. The statistical techniques applied will include a comprehensive method encompassing sociodemographic information, physical activity levels, perceptions of physical literacy, and life satisfaction. The camp shifts were randomly distributed, with half in the control group and the other half in the experimental group . Two measures of physical literacy and life satisfaction were measured: one at the beginning of the camp and one on the day of completion. The intervention included 24 sessions of adventure activities carried out in a natural environment, and the values obtained for both variables were collected using two questionnaires validated for these age groups. This intervention is expected to improve levels of physical literacy and perceived life satisfaction by providing valuable

ELIGIBILITY:
Inclusion Criteria:

* Parental consent
* Participation on summer camps

Exclusion Criteria:

* Older than 18 years
* Not having parental consent.

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 728 (Estimated)
Dates: Start 2025-04-28 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Physical literacy | From day 1 of the camp to day 12 (last day of camp)
  Physical literacy encomprises physical competence, knowledge and understanding and self-expression. This outcome will be assessed by "Students Perceived Physical Literacy Scale", validated by López-Gil et al. (2023) on adolescents. This scale is measured on a 1--5 Likert scale (from 1 "strongly disagree" to 5 "Strongly agree")
Life Satisfaction | From day 1 of camp to 12 days (last day of camp)
  Life satisfaction measure quality of life within last four weeks, according to self perception. This variable will be evaluated by "Students Life Satisfaction Scale", validated on adolescents.

CONTACTS AND LOCATIONS:
Overall Officials: Mayordomo-Pinilla, PhD Student, Principal Investigator — University of Extremadura
Locations (1):
- Sports Science Faculty, Cáceres, Cáceres, Spain

IPD SHARING:
Plan to Share IPD: No